CLINICAL TRIAL: NCT00449696
Title: A Multi-Center, Randomized, Double-Blind, Controlled, Parallel-Group Study of a Single Intra-Articular Injection of Gel-200 With a Single Intra-Articular Injection of Phosphate Buffered Saline (PBS) in Osteoarthritis of the Knee.
Brief Title: Gel-200 Versus Placebo in Osteoarthritis of the Knee
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seikagaku Corporation (Industry)
Responsible Party: Osamu Akahane, Seikagaku Corporation
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SI-6606/01
Record Dates: First submitted 2007-03-20; First posted 2007-03-21 (Estimated); Results first posted 2011-09-15 (Estimated); Last update posted 2011-10-07 (Estimated); Status verified 2011-10

CONDITIONS: Osteoarthritis of the Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gel-200 (Experimental)
  Interventions: Device: Gel-200
- PBS (Placebo Comparator)
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Gel-200 — Single intra-articular injection
  Arms: Gel-200
Device: Placebo — Single intra-articular injection
  Arms: PBS

SUMMARY:
The purpose of this study is to determine if a single intra-articular injection of Gel-200 is superior to a single injection of Phosphate Buffered Saline (PBS) in subjects with symptomatic osteoarthritis of the knee.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a diagnosis of painful, symptomatic tibio-femoral osteoarthritis of the knee (Grade 1-3 on Kellgren - Lawrence (K-L) score).

Exclusion Criteria:

* Subjects with Grade 4 on K-L score
* Subjects with inflammatory diseases of the knee other than osteoarthritis such as rheumatoid arthritis
* Serious systemic diseases
* Female subjects who are pregnant or lactating

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 379 (Actual)
Dates: Start 2006-09; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- SKK, Plantation, Florida, United States

REFERENCES:
- [Derived] Takamura J, Seo T, Strand V. A Pooled Analysis of Two Multicenter, Randomized Controlled Trials of a Single Intra-articular Injection of Gel-200 for Treatment of Osteoarthritis of the Knee. Clin Med Insights Arthritis Musculoskelet Disord. 2018 May 9;11:1179544118773068. doi: 10.1177/1179544118773068. eCollection 2018. PMID 29780263
- [Derived] Strand V, Lim S, Takamura J. Evidence for safety of retreatment with a single intra-articular injection of Gel-200 for treatment of osteoarthritis of the knee from the double-blind pivotal and open-label retreatment clinical trials. BMC Musculoskelet Disord. 2016 Jun 1;17:240. doi: 10.1186/s12891-016-1101-0. PMID 27250845
- [Derived] Strand V, Baraf HSB, Lavin PT, Lim S, Hosokawa H. A multicenter, randomized controlled trial comparing a single intra-articular injection of Gel-200, a new cross-linked formulation of hyaluronic acid, to phosphate buffered saline for treatment of osteoarthritis of the knee. Osteoarthritis Cartilage. 2012 May;20(5):350-356. doi: 10.1016/j.joca.2012.01.013. Epub 2012 Feb 1. PMID 22342928

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 598 patients were screened.
Groups:
- Gel-200: Patients received 1 single dose of Gel-200 (3mL) intra-articular injection into knee joint.
- PBS Placebo: Patients received 1 single dose of Phosphate Buffered Saline (PBS) placebo (3mL) intra-articular injection into knee joint.
Period: Overall Study
Arm/Group | Gel-200 | PBS Placebo
Started | 251 | 128
Received Injection | 249 | 128
Analyzed Participants | 247 (2 subjects removed from ITT analyses because of no post treatment data (pre-defined criteria).) | 128
Completed | 231 | 119
Not Completed | 20 | 9
Not completed — Other Treatment Required | 6 | 1
Not completed — Withdrawal by Subject | 5 | 5
Not completed — Lost to Follow-up | 2 | 3
Not completed — Others | 7 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gel-200 | PBS Placebo | Total
Number analyzed (Participants) | 247 | 128 | 375
Age Continuous [Mean (Standard Deviation); unit: years] | 60.9 (10.24) | 60.3 (9.97) | 60.7 (10.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 147 | 77 | 224
  Male | 100 | 51 | 151
Region of Enrollment [Number; unit: participants]
  United States | 247 | 128 | 375
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms/meters square] | 28.3 (4.14) | 28.7 (3.83) | 28.5 (4.04)
WOMAC VAS Pain Subscore [Mean (Standard Deviation); unit: scores on a scale] — Assessed Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Visual Analog Scale (VAS) pain subscores on VAS of 100 mm.; 0 mm meaning no pain; 100 mm meaning extreme pain.
  scores on a scale | 70.7 (14.42) | 68.0 (13.05) | 69.8 (14.01)
WOMAC VAS Stiffness Subscore [Mean (Standard Deviation); unit: scores on a scale] — Assessed Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Visual Analog Scale (VAS) stiffness subscores on VAS of 100 mm.; 0 mm meaning no stiffness; 100 mm meaning extreme stiffness.
  scores on a scale | 71.6 (17.48) | 69.3 (17.31) | 70.8 (17.43)
WOMAC VAS Physical Function Subcore [Mean (Standard Deviation); unit: scores on a scale] — Assessed Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Visual Analog Scale (VAS) physical function subscores on VAS of 100 mm.; 0 mm meaning no difficulty; 100 mm meaning extreme difficulty.
  scores on a scale | 68.9 (17.41) | 67.6 (15.80) | 68.5 (16.87)
WOMAC VAS Total Score [Mean (Standard Deviation); unit: scores on a scale] — Mean of Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Visual Analog Scale (VAS) pain, stiffness and physical function subscores on VAS of 100 mm.; 0 mm meaning no pain, stiffness and difficulty; 100 mm meaning extreme pain, stiffness and difficulty.
  scores on a scale | 69.5 (15.99) | 67.8 (14.68) | 68.9 (15.56)
Subject Global Evaluations [Mean (Standard Deviation); unit: scores on a scale] — Observed subject evaluations on Visual Analog Scale (VAS) of 100 mm.; 0 mm meaning excellent feeling in knee joint; 100 mm meaning poor feeling in knee joint.
  scores on a scale | 64.7 (21.83) | 66.5 (21.21) | 65.3 (21.61)
Physician Global Evaluations [Mean (Standard Deviation); unit: scores on a scale] — Observed physician evaluations on Visual Analog Scale (VAS) of 100 mm.; 0 mm meaning excellent feeling in knee joint; 100 mm meaning poor feeling in knee joint.
  scores on a scale | 61.5 (14.79) | 64.2 (14.25) | 62.4 (14.65)

OUTCOME MEASURES:

1. Secondary Outcome: Change From Baseline in WOMAC VAS Stiffness Subscore
Description: Observed WOMAC stiffness subscore on Visual Analog Scale (VAS) of 100 mm; 0 mm meaning no stiffness; 100 mm meaning extreme stiffness. Change in score from baseline to week 13 was calculated as baseline minus week 13. Primary endpoint was the model estimated difference between Gel-200 and PBS placebo.
Time Frame: Baseline and Week 13
Population: ITT population was used for analysis. 2 patients with Gel-200 were removed from ITT population analysis and baseline because of no post treatment data according to a pre-specified rule. These data were submitted to FDA.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Gel-200 | PBS Placebo
Number analyzed (Participants) | 247 | 128
scores on a scale | 26.9 (30.46) | 22.5 (28.66)
Statistical Analysis 1: Comparison: Gel-200 vs PBS Placebo; Test type: Superiority or Other; p = 0.122, Quadratic Spline Model; Mean Difference (Net) = 4.91 — Tested superiority of Gel-200 using quadratic spline model for difference between Gel-200 and PBS placebo. Only difference between groups was presented by the pre-specified model as primary endpoint

2. Secondary Outcome: Change From Baseline in WOMAC VAS Physical Function Subscore
Description: Observed WOMAC physical function subscore on Visual Analog Scale (VAS) of 100 mm; 0 mm meaning no difficulty; 100 mm meaning extreme difficulty. Change in score from baseline to week 13 was calculated as baseline minus week 13. Primary endpoint was the model estimated difference between Gel-200 and PBS placebo.
Time Frame: Baseline and Week 13
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Gel-200 | PBS Placebo
Number analyzed (Participants) | 247 | 128
scores on a scale | 26.2 (28.81) | 21.0 (28.62)
Statistical Analysis 1: Comparison: Gel-200 vs PBS Placebo; Test type: Superiority or Other; p = 0.071, Quadratic Spline Model; Mean Difference (Net) = 5.42 — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Change From Baseline in WOMAC VAS Total Score
Description: Mean of all WOMAC pain, stiffness and physical function subscores on Visual Analog Scale (VAS) of 100 mm; 0 mm meaning no pain, stiffness and difficulty; 100 mm meaning extreme pain, stiffness and difficulty. Change in score from baseline to week 13 was calculated as baseline minus week 13. Primary endpoint was the model estimated difference between Gel-200 and PBS placebo.
Time Frame: Baseline and Week 13
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Gel-200 | PBS Placebo
Number analyzed (Participants) | 247 | 128
scores on a scale | 26.6 (28.41) | 21.5 (28.37)
Statistical Analysis 1: Comparison: Gel-200 vs PBS Placebo; Test type: Superiority or Other; p = 0.058, Quadratic Spline Model; Mean Difference (Net) = 5.64 — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Outcome Measures in Rheumatology Arthritis Clinical Trials (OMERACT)- and the Osteoarthritis Research Society International (OARSI) Response
Description: Outcome Measures in Rheumatology Clinical Trials and Osteoarthritis Research Society International (OMERACT-OARSI) strict responses defined by changes from baseline in WOMAC pain or physical function subscore ≥50% with absolute changes ≥20 mm (termed strict responders), or ≥20% with absolute changes ≥10mm in 2 of 3 measures of WOMAC pain or physical function subscore or subject global evaluations (termed responders).
Time Frame: Weeks 6 to 13
Population: as for outcome 1
Measure: Number; unit: Percentage
Arm/Group | Gel-200 | PBS Placebo
Number analyzed (Participants) | 247 | 128
Percentage
  Participants who met strict responders at Week 13 | 45.9 | 38.7
  Participants who met responders at Week 13 | 61.0 | 54.6
Statistical Analysis 1: Comparison: Gel-200 vs PBS Placebo; Test type: Superiority or Other; p = 0.022, Generalized Estimating Equation Model — P-value for strict OMERACT-OARSI response; Odds Ratio (OR) = 1.59
Statistical Analysis 2: Comparison: Gel-200 vs PBS Placebo; Test type: Superiority or Other; p = 0.242, Generalized Estimating Equation Model — P-value for OMERACT-OARSI response; Odds Ratio (OR) = 1.27

5. Secondary Outcome: Change From Baseline in Short Form - 36 (SF-36)
Description: Scored on physical component scale from 0 (negative health) to 100 (positive health). Calculated norm based with a mean of 50 and a standard deviation of 10.
Time Frame: Baseline and Week 13
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores
Arm/Group | Gel-200 | PBS Placebo
Number analyzed (Participants) | 247 | 128
scores | 4.6 (9.34) | 5.3 (9.04)
Statistical Analysis 1: Comparison: Gel-200 vs PBS Placebo; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney) — P-value for physical component scores, physical function subscale, role physical subscale, and bodily pain subscale

6. Primary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Visual Analog Scale (VAS) Pain Subscore
Description: Observed WOMAC pain subscore on VAS of 100 mm; 0 mm meaning no pain; 100 mm meaning extreme pain. Change in score from baseline to week 13 was calculated as baseline minus week 13. Primary endpoint was the model estimated difference between Gel-200 and PBS placebo.
Time Frame: Baseline and Week 13
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Gel-200 | PBS Placebo
Number analyzed (Participants) | 247 | 128
scores on a scale | 27.8 (29.26) | 22.6 (29.31)
Statistical Analysis 1: Comparison: Gel-200 vs PBS Placebo; Test type: Superiority or Other; p = 0.037, Quadratic Spline Model; Mean Difference (Net) = 6.39 — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Change From Baseline in Subject Global Evaluations
Description: Observed subject evaluations on Visual Analog Scale (VAS) of 100 mm; 0 mm meaning excellent feeling in knee joint; 100 mm meaning poor feeling in knee joint. Change in score from baseline to week 13 was calculated as baseline minus week 13. Primary endpoint was the model estimated difference between Gel-200 and PBS placebo.
Time Frame: Baseline and Week 13
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Gel-200 | PBS Placebo
Number analyzed (Participants) | 247 | 128
scores on a scale | 22.8 (33.08) | 22.0 (30.58)
Statistical Analysis 1: Comparison: Gel-200 vs PBS Placebo; Test type: Superiority or Other; p = 0.746, Quadratic Spline Model; Mean Difference (Net) = 0.92 — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Change From Baseline in Physician Global Evaluations
Description: Observed physician global evaluations on Visual Analog Scale (VAS) of 100 mm; 0 mm meaning excellent feeling in knee joint; 100 mm meaning poor feeling in knee joint. Change in score from baseline to week 13 was calculated as baseline minus week 13. Primary endpoint was the model estimated difference between Gel-200 and PBS placebo.
Time Frame: Baseline and Week 13
Population: ITT population was used for analysis. 2 patients with Gel-200 were removed from ITT population analysis and baseline because of no post treatment data according to a pre-specified rule.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Gel-200 | PBS Placebo
Number analyzed (Participants) | 247 | 128
scores on a scale | 21.3 (28.46) | 19.0 (26.97)
Statistical Analysis 1: Comparison: Gel-200 vs PBS Placebo; Test type: Superiority or Other; p = 0.166, Quadratic Spline Model; Mean Difference (Net) = 3.56 — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Acetaminophen Consumption
Description: Weekly mean acetaminophen consumption between weeks 9 and 13.
Time Frame: Weeks 9 to 13 (5 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Gel-200 | PBS Placebo
Number analyzed (Participants) | 247 | 128
milligrams | 2007 (3687) | 2599 (3806)
Statistical Analysis 1: Comparison: Gel-200 vs PBS Placebo; Test type: Superiority or Other; p = 0.041, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Gel-200 | PBS Placebo
Serious Adverse Events (participants affected / at risk) | 8/249 | 0/128
Other Adverse Events (participants affected / at risk) | 122/249 | 55/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gel-200 (N=249) | PBS Placebo (N=128)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 0 (0)
Femoral hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cryptogenic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Transient Ischemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Exertional Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gel-200 (N=249) | PBS Placebo (N=128)
Upper respiratory tract infections (Infections and infestations) | 16 (16) | 6 (6)
Joint swelling (Musculoskeletal and connective tissue disorders) | 70 (91) | 36 (42)
Joint effusion (Musculoskeletal and connective tissue disorders) | 58 (69) | 33 (40)
Arthralgia (Musculoskeletal and connective tissue disorders) | 44 (55) | 15 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
SKK has the right to review the disclosures. Investigator shall not make any publication of study data, information, results or similar information without the express of permission of SKK.